CLINICAL TRIAL: NCT00337233
Title: Restorative Yoga for Symptom Management and Stress Reduction in Women With Ovarian Cancer
Brief Title: Yoga in Controlling Symptoms and Reducing Stress in Women With Ovarian Cancer or Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000481279; CCCWFU-02403; CCCWFU-BG03-658
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2015-09

CONDITIONS: Breast Cancer; Fatigue; Ovarian Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: fatigue; psychosocial effects of cancer and its treatment; recurrent breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian epithelial cancer; stage I ovarian germ cell tumor; stage II ovarian epithelial cancer; stage II ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: yoga therapy — 10 week yoga class

SUMMARY:
RATIONALE: Yoga may improve symptoms and quality of life and reduce stress in patients with ovarian cancer or breast cancer and may help them live more comfortably.

PURPOSE: This clinical trial is studying how well yoga works in controlling symptoms and reducing stress in women with ovarian cancer or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of implementing a restorative yoga intervention as a complementary supportive therapy for women with ovarian or breast cancer.
* Measure changes in fatigue, psychosocial distress (anxiety, depression), psychological well-being (positive emotions), and overall quality of life from baseline to completion of the study treatment.

OUTLINE: This is a pilot study.

Patients undergo a 75-minute restorative yoga session once a week for 10 weeks.

Patients complete questionnaires regarding fatigue, psychological distress (anxiety, depression), positive affect, and quality of life at baseline, immediately after the final yoga session, and then at 2 months after the final yoga session.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast or ovarian cancer

  * Must be 2-24 months post-primary treatment (e.g., surgery) for breast cancer and/or have had a recurrence of breast cancer within the past 24 months
  * Must be 3-24 months post-primary treatment (e.g., surgery) for ovarian cancer and/or have had a recurrence of ovarian cancer within the past 24 months
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Female
* Menopausal status not specified
* Zubrod performance status 0-3
* No medical contraindications
* Understands written and spoken English

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2004-01; Primary Completion 2006-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Fatigue as measured by the FACT-Fatigue subscale | 18 weeks
Psychological distress as measured by the Center for Epidemiologic Studies-Depression Scale and the State-Trait Anxiety Inventory | 18 weeks
Positive affect as measured by the Positive and Negative Affect Schedule | 18 weeks
Quality of life as measured by Functional Assessment of Cancer Therapy (FACT-O) for patients with ovarian cancer or FACT-B for patients with breast cancer | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne C. Danhauer, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Danhauer SC, Mihalko SL, Russell GB, Campbell CR, Felder L, Daley K, Levine EA. Restorative yoga for women with breast cancer: findings from a randomized pilot study. Psychooncology. 2009 Apr;18(4):360-8. doi: 10.1002/pon.1503. PMID 19242916